CLINICAL TRIAL: NCT04320576
Title: Long-term Clinical Comparison of Bulk-fill and Nano-fill Composite Restorations
Brief Title: Clinical Comparison of Bulk-fill Restorative and Nano-fill Resin Composite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zeynep Bilge Kutuk, Assistant Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04(KA-15004)
Record Dates: First submitted 2020-03-22; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bulk-fill resin composite (Experimental): Bulk-fill resin composite will be places with bulk technique.
  Interventions: Device: Bulk-fill
- Nano-fill resin composite (Active Comparator): Nano-fill resin composite will be placed with 2 mm thickness layering technique.
  Interventions: Device: Nano-fill

INTERVENTIONS:
Device: Bulk-fill — Bulk-fill resin composite (bulk technique)
  Arms: Bulk-fill resin composite
Device: Nano-fill — Nano-fill resin composite (layering technique)
  Arms: Nano-fill resin composite

SUMMARY:
The aim of this study is to evaluate the clinical performance of a nano-fill and a bulk fill resin composite in class II restorations.

DETAILED DESCRIPTION:
In accordance with a split-mouth design, 50 patients will be received at least one pair of restorations, restored with a nanofill resin composite (Filtek Ultimate [FU]) and with a bulk fill resin composite (Tetric EvoCeram Bulk Fill [TB]). Each restorative resin will be used with its respective adhesive system according to the manufacturers' instructions. A total of 104 class II restorations will be placed by two operators. The restorations will be blindly evaluated by two examiners at baseline and at 1-, 2-, 3-, 4-, 5-, 6-, 7- and 8- year using modified US Public Health Service Ryge criteria. The comparison of the two restorative materials for each category will be performed with the chi-square test (a=0.05). The baseline scores will be compared with those at the recall visits using the Cochran Q-test.

ELIGIBILITY:
Inclusion Criteria:

* a need for at least two but not more than four posterior tooth-colored restorations
* the presence of teeth to be restored in occlusion
* teeth that were symptomless and vital
* a normal periodontal status
* a good likelihood of recall availability.

Exclusion Criteria:

* partly erupted teeth
* absence of adjacent and antagonist teeth
* poor periodontal status
* adverse medical history
* potential behavioral problems

Ages: 24 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-05-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Marginal adaptation | From baseline to 8 year the change of restorations will be evaluated
  Observers will evaluate the restorations will be performed using the modified United State Public Health Service criteria regarding marginal adaptation.
  Marginal adaptation will evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches will be performed . A score means the higher score of clinical acceptability while C and D score means that the restoration has failed and needs to be replaced. Alpha 1: Harmonious outline Alpha 2: Marginal gap (max 100μ) with discoloration (removable) Bravo: Marginal gap (> 100μ) with discoloration (unremovable) Charlie: The restoration is fractured or missed.
Marginal discoloration | From baseline to 8 year the change of restorations will be evaluated
  Observers will evaluate the restorations will be performed using the modified United State Public Health Service criteria regarding marginal discoloration.
  Marginal discoloration will be evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches will be performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth. Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth. Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction.
Retention | From baseline to 8 year the change of restorations will be evaluated
  Observers will evaluate the restorations will be performed using the modified United State Public Health Service criteria regarding retention rate.
  Retention rate will be evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C and D score means that the restoration has failed and needs to be replaced. Alpha 1:Clinically excellent Alpha 2: Clinically good with slight deviations from ideal performance, correction possible without damage of tooth or restoration Bravo: Clinically sufficient with few defects, corrections or repair of the restoration possible Charlie: Restoration is partially missed Delta: Restoration is totally missed
Anatomic form | From baseline to 8 year the change of restorations will be evaluated
  Observers will evaluate the restorations will be performed using the modified United State Public Health Service criteria regarding anatomic form.
  Anatomic form will be evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha 1: Continuous with existing anatomical form Alpha 2: Slightly discontinuous due to some chipping on the proximal ridge Bravo: Discontinuous with existing anatomical form due to material loss but proximal contact still present Charlie: Proximal contact is lost with ridge fracture.
Color change | From baseline to 8 year the change of restorations will be evaluated
  Observers will evaluate the restorations will be performed using the modified United State Public Health Service criteria regarding color change. Color changes will be evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failedand needs to be replaced. Alpha: The restoration matches the adjacent tooth structure in color and translucency. Bravo: Light mismatch in color, shade or translucency between the restoration and the adjacent tooth. Charlie: The mismatch in color and translucency is outside the acceptable range of tooth color and translucency.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse R Yazici, DDS, PhD, Study Director — Hacettepe University School of Dentistry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PUBMED — https://www.ncbi.nlm.nih.gov/pubmed/28581919
- See also: PUBMED — https://www.ncbi.nlm.nih.gov/pubmed/29630489